CLINICAL TRIAL: NCT03807466
Title: Feedback to Improve Rational Strategies of Antibiotic Initiation and Duration in Long Term
Brief Title: Feedback to Improve Rational Strategies of Antibiotic Initiation and Duration in Long Term Care
Acronym: FIRST AID-LTC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Clinical Evaluative Sciences (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Agency for Health Protection and Promotion (Other Government); Health Quality Ontario (Other)
Responsible Party: Principal Investigator, Nick Daneman, Adjunct Scientist, Institute for Clinical Evaluative Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 441-2017
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Antibiotic Initiation; Antibiotic Duration

STUDY DESIGN:
Intervention Model Description: Assess two interventional parallel study models consisting of two intervention arms each
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The team at Health Quality Ontario will be aware of the physicians' assignment to dynamic versus paginated reports so that they can send the correct audit-and-feedback document. However, the analytic team at ICES will be masked, and outcome data will be extracted by the analysis team from routinely collected administrative databases (Ontario drug benefits database).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dynamic/Interactive Report (Active Comparator): LTC physician receives dynamic/interactive report only
  Interventions: Behavioral: Dynamic/Interactive vs. Static/Paginated Report
- Static/Paginated Report (No Intervention): LTC physician receives static/paginated report only
- LTC Physicians Enrolled in Reports (Active Comparator): All LTC physicians who receive a dynamic or paginated report
  [note: this is not part of randomization assignment, but a quasi-experimental study]
  Interventions: Behavioral: LTC Physicians Enrolled vs. Not Enrolled in Reports
- LTC Physicians Not Enrolled in Reports (No Intervention): All LTC physicians who do not receive a dynamic or paginated report
  [note: this is not part of randomization assignment, but a quasi-experimental study]

INTERVENTIONS:
Behavioral: Dynamic/Interactive vs. Static/Paginated Report — Evaluate whether a stand-alone interactive audit-and-feedback report highlighting antibiotic prescribing can lead to greater reductions in antibiotic use, than a report embedded in a broader static feedback system
  Arms: Dynamic/Interactive Report
Behavioral: LTC Physicians Enrolled vs. Not Enrolled in Reports — Evaluate whether being provided an audit-and-feedback report (regardless of dynamic or static) can lead to greater reductions in antibiotic use, than those who do not receive either report
  Arms: LTC Physicians Enrolled in Reports

SUMMARY:
There is a high rate of inappropriate antibiotic use in long-term care (LTC) facilities, with both unnecessary initiation and prolongation of treatments. Although there are challenges to rational antibiotic use in LTC, the variability in antibiotic initiation and use of prolonged treatment durations is driven by prescriber tendencies rather than resident characteristics. Audit-and-feedback is a well-established intervention to improve professional practices, and is ideally suited for use to improve antibiotic prescribing tendencies in LTC. The literature is saturated with trials indicating benefit of audit-and-feedback, but is in dire need of studies to identify methods to improve the impact of this technique. Health Quality Ontario (HQO), a key partner in the FIRST AID-LTC research program, is already providing audit-and-feedback for other inappropriate prescribing practices in LTC, and has identified antibiotic prescribing as a priority focus.

DETAILED DESCRIPTION:
Overarching Goals

The overarching goals of FIRST AID - LTC are two-fold:

1. Improve rational antibiotic prescribing by physicians to minimize harms among LTC residents.
2. Advance the science of audit-and-feedback to improve physician prescribing practices.

Specific Aims

To improve rational antibiotic prescribing in LTC:

1. by decreasing unnecessary initiation of antibiotic treatments among Ontario LTC residents, as well as the variability in initiation rates across LTC prescribers.
2. by decreasing unnecessary prolonged duration of antibiotic treatments among Ontario LTC residents, as well as the variability in prolonged duration treatment use across LTC prescribers.

To advance audit-and-feedback implementation science:

1. by evaluating whether a dynamic audit-and-feedback report highlighting antibiotic prescribing can lead to greater reductions in antibiotic use, than a static paginated report

Anticipated Contributions to Health-Related Knowledge

Although the literature is inundated with trials examining the impact of audit-and-feedback compared to usual care, there is a need for studies to improve audit-and-feedback delivery. FIRST AID-LTC will test optimal delivery and peer comparison techniques for audit-and-feedback. The knowledge learned can be extrapolated to antibiotic interventions in LTC in other provinces across Canada, as well more broadly to inappropriate medication prescribing practices in LTC.

Anticipated Contributions to Health Care, Health Systems and Health Outcomes

FIRST AID-LTC will lead to immediate reductions in excess antibiotic use in Ontario LTC facilities, which in turn should result in substantial reductions in direct drug costs, as well as downstream complications of allergy, organ toxicity, C. difficile infections and antimicrobial resistance. With easy transferability to other Canadian provinces, the improvements in cost-savings and patient outcomes could be massive in scope.

ELIGIBILITY:
To Identify an LTC Resident

Inclusion Criteria:

An individual having a minimum of 2 records on separate days within the quarter meeting any combination of the following criteria:

* a record for a non-emergency long-term care inpatient services OR
* an Ontario Drug Benefits record administered in long-term care

Index date = The analysis will be anchored on the most recent of either of the records above within a given quarter or their date of death (whichever date is earliest)

Exclusion Criteria:

* Non-Ontario resident at index date
* Invalid age (age<19 or age>115) at index date
* Missing or invalid sex or date of birth at index date
* Death date is >7 days before index date
* If the individual does not live in a nursing home or home for the aged
* Cannot be linked to a Most Responsible Physician (MRP) (see methodology below)

To Identify the Most Responsible Physician (MRP) Using Virtual Rostering

For each patient in the above resident cohort, the study team will retrieve all records from health care providers in the 6 month period preceding the index date (180 days), keeping only records from physicians who have a specialty of 1) general practice, 2) community medicine or 3) geriatrics.

Steps for MRP assignment:

Step 1) The study team will first select physicians with the highest count of records for the monthly management of a nursing home or home for the aged. This is completed for as many residents as possible.

Step 2) If there were no monthly management fee records as described above then the physician with highest count of non-emergency long-term care inpatient services records for each patient will be selected. This step is only applied to residents who could not be matched to a physician by Step 1. **Physician must have seen the patient one or more times in 90 days prior to and including index date to be considered MRP. This criteria is applied to ensure the physician has seen the resident within the reporting quarter.

Step 3) Some patients will virtually roster to physicians in Enrollment groups, some will virtually roster to physicians that are not in a group. For these, the study team will recode enrollment program type to 'NOR' (not otherwise rostered) - these are likely fee for service physicians.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Antibiotic initiation | 3 months
  Median % of patients initiated on an antibiotic
Antibiotic duration | 3 months
  Median % of antibiotic treatments prolonged >7 days

SECONDARY OUTCOMES:
ER visit or hospitalization for infection | 3 months
  The percentage of a LTC physicians' patients that experienced an ER visit or hospitalization due to a potential antibiotic-related harm, including: allergy, general medication adverse event, diarrhea, C. difficile infection, or infection with an antibiotic-resistant organism
ER visit or hospitalization for antibiotic harms | 3 months
  To test for harms related to decreased antibiotic use by comparing the percentage of LTC physicians' patients that experience an infection-related ER visit or admission
Net Clinical impact | 3 months
  Measure the net clinical impact of the intervention, by comparing all-cause ER visits and hospitalizations and mortality
Anti-psychotic use | 3 months
  The percent reduction in anti-psychotic use
Benzodiazepine use | 3 months
  The percent reduction in benzodiazepines

CONTACTS AND LOCATIONS:
Overall Officials: Nick Daneman, MD, Principal Investigator — ICES
Locations (1):
- ICES, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daneman N, Lee SM, Bai H, Bell CM, Bronskill SE, Campitelli MA, Dobell G, Fu L, Garber G, Ivers N, Lam JMC, Langford BJ, Laur C, Morris A, Mulhall C, Pinto R, Saxena FE, Schwartz KL, Brown KA. Population-Wide Peer Comparison Audit and Feedback to Reduce Antibiotic Initiation and Duration in Long-Term Care Facilities with Embedded Randomized Controlled Trial. Clin Infect Dis. 2021 Sep 15;73(6):e1296-e1304. doi: 10.1093/cid/ciab256. PMID 33754632
- [Derived] Laur C, Sribaskaran T, Simeoni M, Desveaux L, Daneman N, Mulhall C, Lam J, Ivers NM. Improving antibiotic initiation and duration prescribing among nursing home physicians using an audit and feedback intervention: a theory-informed qualitative analysis. BMJ Open Qual. 2021 Feb;10(1):e001088. doi: 10.1136/bmjoq-2020-001088. PMID 33547157